CLINICAL TRIAL: NCT00629720
Title: Four-week, Open-label, Multicenter, Randomized, Parallel-group Study to Investigate the Pharmacokinetics, Safety, Tolerability and the Effects on Leak Point Pressure of Two Oral Doses of Alfuzosin (0.1 mg/kg/Day; 0.2 mg/kg/Day) in Children and Adolescents 2 to 16 Years-of-age With Elevated Detrusor Leak-point Pressure of Neuropathic Etiology
Brief Title: Pharmacokinetics and Safety Study With Alfuzosin in Children and Adolescents With Elevated Detrusor Leak Point Pressure of Neuropathic Etiology
Acronym: ALFACHIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKM6270
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Urinary Bladder Neurogenic
Keywords: elevated detrusor leak point pressure
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — alfuzosin

INTERVENTIONS:
Drug: alfuzosin (SL770499)

SUMMARY:
The primary objective is to investigate the pharmacokinetics (PK) of 2 doses of alfuzosin (given as a solution or tablets depending on age) in children and adolescents 2 to 16 years of age with elevated detrusor Leak Point Pressure (LPP) (≥40 cm H2O) of neuropathic etiology stratified into 2 age groups (2 to 7 years and 8 to 16 years).

The secondary objectives are to investigate the safety and tolerability of the 2 dose regimens and to determine the effect of the 2 dose regimens on detrusor LPP.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents of either gender 2-16 years of age with elevated detrusor LPP of neuropathic etiology.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2006-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
PK parameters

SECONDARY OUTCOMES:
Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Malvern, Pennsylvania, United States
- Sanofi-Aventis Administrative Office, Belgrade, Serbia